CLINICAL TRIAL: NCT03384069
Title: Cognitive Behavioral Therapy for African Americans With Mild Cognitive Impairment
Brief Title: CBT for African Americans With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Ambar Kulshreshtha, Asstant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00099440
Record Dates: First submitted 2017-12-13; First posted 2017-12-27 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease
Keywords: Cognitive Impairment; Cognitive- behavioral therapy; African Americans
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-based Cognitive Behavioral Therapy (CBT) (Experimental): The Group-based CBT will incorporate psycho-education about cognitive behavioral skills and written materials to support learning and application of the psycho-educational content. The intervention will be culturally tailored to incorporate beliefs/attitudes, health literacy, effective communication, and motivational strategies, which focus on African Americans.
  Interventions: Behavioral: Group-based Cognitive Behavioral Therapy (CBT)
- Phone-based Cognitive Behavioral Therapy (CBT) (Experimental): This intervention will follow the same protocol as the group-based CBT, but without the opportunity for group-interaction. It will incorporate psycho-education about cognitive behavioral skills and written materials to support learning and application of the psycho-educational content. The intervention will be culturally tailored to incorporate beliefs/attitudes, health literacy, effective communication, and motivational strategies, which focus on African Americans.
  Interventions: Behavioral: Phone-based Cognitive Behavioral Therapy (CBT)
- Standard of care (No Intervention): Participants will continue to receive care and follow up from their primary care providers, that incorporates general education regarding lifestyle activities and AD prevention.

INTERVENTIONS:
Behavioral: Group-based Cognitive Behavioral Therapy (CBT) — The group-based CBT intervention will include twelve 1-hour group sessions held biweekly for six months. Each sixty-minute session will consist of 15 minutes of Alzheimer's disease (AD) prevention education and approximately 45 minutes of CBT presentations/engagement activities. A physician and a Behavioral Interventionist will collaboratively facilitate the group sessions.
  Arms: Group-based Cognitive Behavioral Therapy (CBT)
Behavioral: Phone-based Cognitive Behavioral Therapy (CBT) — Participants in the phone-based CBT will be asked to reserve a 1-hour period for a phone call from the Behavioral Interventionist biweekly for six months. Text reminders will be sent to the participant's prior the sessions. This intervention will follow the same frequency and format as the group-based CBT and will use an established protocol incorporating the same elements of cognitive behavior change as in the group-based CBT, but without the opportunity for group-interaction.
  Arms: Phone-based Cognitive Behavioral Therapy (CBT)

SUMMARY:
The aim of the study is to test the feasibility and acceptability of a six-month cognitive-behavioral therapy (CBT) program (group based and phone-based) compared with usual care, and to determine if the intervention can improve cognitive performance and reduce chronic stress in a randomized trial including 30 African American patients with Mild Cognitive Impairment (MCI). The CBT program among African Americans with MCI will provide preliminary evidence about the efficacy and the optimal intensity of the intervention needed for patients at risk of Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) can involve problems with memory, language, thinking and judgment that are greater than normal age-related changes and it maybe a precursor for Alzheimer's disease. African Americans have a higher risk of developing MCI compared with Whites. Unfortunately, prevention and management of MCI has been understudied among African-Americans. Chronic stress (such as perceived discrimination, daily environmental stress) in African Americans can affect cognition and also plays a role in worsening of unhealthy behaviors such as smoking, improper diet and physical inactivity. Cognitive-behavioral therapy (CBT) is a collaborative psychological approach that addresses the interaction between people's thoughts, feelings and behavior. Existing evidence suggests that CBT can be an effective strategy for dementia patients with co-morbid anxiety. However, none of these studies have specifically evaluated African Americans with MCI. The aim of the study is to test the feasibility and acceptability of a six-month CBT program (group based and phone-based) compared with usual care, and to determine if the intervention can improve cognitive performance and reduce chronic stress in a randomized trial including 30 African American patients with MCI. The CBT program among African Americans with MCI will provide preliminary evidence about the efficacy and the optimal intensity of the intervention needed for patients at risk of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 years or older
* Race: African American
* Fluency in English
* Mild Cognitive Impairment (MCI) - defined as subjective memory complaints with a Montreal Cognitive Assessment (MoCA) 18- 26

Exclusion Criteria:

* Dementia diagnosis or reversible causes of dementia (e.g. if the patient has hypothyroidism or low vitamin B12 that is contributing to the subject's cognitive impairment)
* Active medical or psychiatric diseases that in the judgment of the investigator would affect the safety of the subject or scientific integrity of the study (e.g. actively manic patient)
* Uncontrolled medical conditions (such as congestive heart failure) reflected by poor exercise tolerance and shortness of breath
* Any physical ailment (such as stroke with residual impairment) that is a barrier to perform study procedures and attend sessions.
* Those who are unable to demonstrate that they understood the details of the study (i.e. lack of decisional- capacity to consent) or linguistic limitations will be excluded;
* Pregnant women
* Prisoners
* Adults unable to consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Number of participants attending CBT sessions (participants retention) | 3 and 6 months follow up
  Participants retention will be estimated by number of participants attending CBT sessions.
Percentage of patients enrolled as per target (feasibility) | Baseline
  Feasibility of the six-month cognitive-behavioral therapy (CBT) program will be estimated by percentage of patients enrolled as per target.

SECONDARY OUTCOMES:
Change in attitudes of patients regarding a CBT intervention for Mild Cognitive Impairment (MCI) | Baseline, 3 and 6 months follow up
  Semi-structured interviews will be used to assess attitudes of patients. The questions in each will be designed to examine attitudes towards the diagnosis of MCI, CBT approach for prevention, effectiveness of the intervention. Trained staff will conduct the focus group interviews, audiotaped (with the permission of participants) and transcribed verbatim. The ATLAS.ti software will be used to retrieve all quotations in a code category for comparison and refinement.
Change in the Center for Epidemiological Studies-Depression (CESD-R) score | Baseline, 3 and 6 months follow up
  The CESD-R is a screening test for depression and depressive disorder. The CESD-R measures symptoms defined by the American Psychiatric Association' Diagnostic and Statistical Manual (DSM-V) for a major depressive episode. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Change in Perceived Stress Scale (PSS) score | Baseline, 3 and 6 months follow up
  The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all 10 scale items.
Change in the quality of life scale (36-Item Short-Form Health Survey (SF-36)) score | Baseline, 3 and 6 months follow up
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ambar Kulshreshtha, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta, Georgia, United States